CLINICAL TRIAL: NCT00672295
Title: A Phase I Trial of A SRC Kinase Inhibitor, Dasatinib,in Combination With Paclitaxel and Carboplatin in Patients With Advanced or Recurrent Ovarian, Peritoneal, and Tubal Cancer
Brief Title: PH I SRC Kinase, Dasatinib Combo Paclitaxel & Carboplatin in Pts w Ovarian, Peritoneal, & Tubal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AA Secord (Other)
Responsible Party: Sponsor-Investigator, AA Secord, Associate Professor, Gynecologic Oncology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00012282; 105821b; 9311-06-R0
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Ovarian Cancer; Peritoneal Cancer; Tubal Cancer; Fallopian Tube Cancer; Dasatinib; Sprycel; Paclitaxel; Taxol; Carboplatin; Paraplatin
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Dasatinib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib, paclitaxel,and carboplatin (Experimental): Combination of dasatinib, paclitaxel,and carboplatin
  Interventions: Drug: Dasatinib, Paclitaxel, and Carboplatin

INTERVENTIONS:
Drug: Dasatinib, Paclitaxel, and Carboplatin — Dasatinib will be administered as an oral dose (tablet) as per the dose escalation (50 mg everyday - 250 mg everyday)continuously on days 2-21 in the first cycle (3 weeks) therapy and continuously (days 1-21) throughout the remainder of therapy.
  Paclitaxel will be administered on a 21-day schedule. Paclitaxel (150-175 mg/m^2) IV infused over 3 hours on day #1 of each cycle.
  Carboplatin (AUC=5-6 mg/,l/min) will be infused over 30-60 minutes every cycle via IV on day 1 of every cycle following the paclitaxel administration.
  All patients will be followed until disease progression or study withdrawal. In addition, following disease progression, patients will be monitored for delayed toxicity and survival for a period of 5 years and data entered into eDC, unless is withdrawn.
  Other Names: Dasatinib; Paclitaxel; Carboplatin; Taxol; Paraplatin; Sprycel

SUMMARY:
Primary objective to determine the maximal tolerated (MTD) of dasatinib in combination with paclitaxel and carboplatin during the first cycle of treatment.

Secondary objectives to describe the toxicity of this combination of therapy; to describe the pharmacokinetics and pharmacodynamics parameters related to this combination; to describe the clinical activity as defined as the response rate (complete and partial response rate) and progression-free survival > 6 month; to compare the SRC pathway microarray signature in pre and post-treatment cancer specimens; to evaluate SRC pathway downstream substrates, FAX, paxcillin, and CRK-L in pre and post-treatment cancer specimens.

DETAILED DESCRIPTION:
This is a phase I multicenter study designed to determine the maximal tolerated dose (MTD) and toxicity of dasatinib in combination with paclitaxel and carboplatin during the first cycle of treatment in patients with advanced or recurrent ovarian, peritoneal, and tubal carcinoma. The MTD will be defined as the highest dose at which no more than 1 of 6 evaluable patient experiences a dose-limiting toxicity (DLT) due to the combination of dasatinib, paclitaxel,and carboplatin during the first cycle of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pts must have histologic or cytologic evidence of ovarian, peritoneal, or tubal cancer
* All pts must have measurable disease
* > 18 yrs
* Expected survival of at least 3 months
* Pts must have GOG performance status pf 0, 1 or 2
* Pts must have adequate:Bone marrow function, renal function, hepatic function, neurologic function
* No chemo, radiotherapy, biologic, hormonal, or investigational drug therapy within 28 days prior to study entry
* Pts may have had up to 3 prior cytotoxic chemo regimens including prior treatment w carboplatin & paclitaxel
* Capable of providing written informed consent
* Pts of childbearing potential must have negative serum pregnancy test prior to study entry & be practicing effective method of birth control during course of study, in manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential must be advised of importance of avoiding pregnancy during trial participation & potential risk factors for unintentional pregnancy
* Pts must have tissue block from their tumor available for evaluation for microarray & immunoblot analyses. Pretreatment tumor tissue may be obtained from either archival tissue or be obtained by guided by guided core needle or simple biopsy it must be performed within four weeks prior to enrollment on study. Pts must have tumor that is accessible to biopsy & consent to undergo post-treatment biopsy after cycle #2 of treatment as well

Exclusion Criteria:

* Pts w epithelial ovarian tumors of low malignant potential (borderline tumor)
* Pts w history of other invasive malignancies, w exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within last 5 yrs
* Pts who have following cardiac conditions: uncontrolled angina or myocardial infarction within past 6 months; diagnosed or suspected congenital long QT syndrome; Any history of clinically significant ventricular arrhythmias; Prolonged QTc interval on pre-entry electrocardiogram on both Fridericia & Bazett's correction; uncontrolled hypertension
* History of significant bleeding disorder unrelated to cancer, including: diagnosed congenital bleeding disorders; diagnosed acquired bleeding disorder within 1 yr
* Pts currently taking drugs that are generally accepted to have risk of causing Torsades de Pointes including: quinidine, procainamide, disopyramide; amiodarone, sotalol, ibutilide, dofetilide; erythromycins, clarithromycin; chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide; cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* Serum creatinine > 1.5 times institutional upper limits of normal
* Pts taking certain concomitant medications, consider following prohibitions: medications that inhibit platelet function or anticoagulants
* Pts who have received radiation therapy to > 30 percent of bone marrow
* Pts w history of grade 3 hypersensitivity to paclitaxel or carboplatin
* Pts w septicemia, severe infection, acute hepatitis, other uncontrolled severe medical conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-08; Primary Completion 2011-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To determine maximal tolerated dose (MTD) of dasatinib in combination with paclitaxel and carboplatin during the first cycle of treatment | 6 months

SECONDARY OUTCOMES:
To describe the toxicity of this combination of therapy | 6 months
To describe the pharmacokinetics and pharmacodynamics parameters related to this combination | 6 months
To describe the clinical activity as defined as the response rate (complete and partial response rate) and progression-free survival > 6 months | 6 months
To compare the SRC pathway microarray signature in pre and post-treatment cancer specimens | 6 months
To evaluate SRC pathway downstream substrates, FAX, paxcillin, and CRK-L in pre and post-treatment cancer specimens | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Angeles A Secord, MD, Principal Investigator — Duke Health
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Duke University Health System, Durham, North Carolina

REFERENCES:
- [Background] Secord AA, Teoh DK, Barry WT, Yu M, Broadwater G, Havrilesky LJ, Lee PS, Berchuck A, Lancaster J, Wenham RM. A phase I trial of dasatinib, an SRC-family kinase inhibitor, in combination with paclitaxel and carboplatin in patients with advanced or recurrent ovarian cancer. Clin Cancer Res. 2012 Oct 1;18(19):5489-98. doi: 10.1158/1078-0432.CCR-12-0507. Epub 2012 Jul 26. PMID 22837181
- See also: Related Info — http://obgyn.duke.edu